CLINICAL TRIAL: NCT00038012
Title: A Pilot Study of Transfusion of rhTPO-Derived Autologous Platelets Cryopreserved With Thrombosol and 2% DMSO in Patients With Gynecologic Malignancy Receiving Carboplatin
Brief Title: rhTPO Mobilized Auto Cryo Platelets For GYN Patients Receiving Carboplatin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pharmacia (Industry); LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYN97-310
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms, Gynecologic
Keywords: Dose-intensified carboplatin; autologous cryopreserved platelets; thrombopoietin; Gynecologic malignancy
MeSH Terms: conditions — Genital Neoplasms, Female; Jacobs syndrome | interventions — Thrombopoietin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rhTPO-Derived Autologous Platelets Transfusion (Experimental)
  Interventions: Drug: Thrombopoietin; Procedure: Platelet-pheresis; Drug: Carboplatin

INTERVENTIONS:
Drug: Thrombopoietin
Procedure: Platelet-pheresis
Drug: Carboplatin
  Other Names: Paraplatin

SUMMARY:
A Pilot Study of Transfusion of rhTPO-Derived Autologous Platelets Cryopreserved with ThromboSol and 2% DMSO in Patients with Gynecologic Malignancy Receiving Carboplatin

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with gynecologic malignancy for whom treatment with carboplatin is indicated.
* Age >/= 15 years.
* Adequate hematologic, renal, and hepatic functions.
* Life expectancy >/- 3 months. Karnofsky Performance Status >/= 80.
* Signed informed consent form.

EXCLUSION CRITERIA:

* Patients with rapidly progressive disease.
* Pregnant or lactating women.
* Patients with comorbid condition which renders patients at high risk of treatment complication.
* History of CNS metastasis.
* Patients with significant cardiac disease (NYHA Class III or IV), dysrhythmia, or recent history of MI or ischemia, transient ischemic attack or CVA within the 6 months of study entry.
* Prior chemotherapy, immunotherapy, any experimental drug within 4 weeks, use of myeloid (G-CSF or GM-CSF) growth factors within 2 weeks or erythropoietin within 4 weeks.
* Use of any nitrosourea (BCNU, CCNU) or mitomycin - C within 6 weeks.
* Prior surgery or RT within 2 wks of study entry.
* Patients with history of prior high dose chemotherapy with stem cell transplant or with history of prolonged thrombocytopenia (> 2 weeks).
* History of leukemia.
* History of any platelet disorders including ITP, TTP or bleeding disorders.
* History of > 3 prior chemotherapy regimens (all platinum regimens will be counted as 1 regimen).
* Demonstrated lack of response to platinum-based therapy.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1999-07-23 (Actual); Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Response Rate | Continuous

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org